CLINICAL TRIAL: NCT00387296
Title: FAST Lidocaine, "Study of Functional Microarray-Facilitated Lidocaine Liposomal Cream Absorption for Cutaneous Anesthesia in Volunteers"
Brief Title: Study of Functional Microarray-Facilitated Lidocaine Liposomal Cream Absorption for Cutaneous Anesthesia in Volunteers
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding nonavailability and principal investigator move
Sponsor: Massachusetts General Hospital (Other)
Collaborators: NanoMed Pharmaceuticals (Industry)
Responsible Party: Stephen H. Thomas MD MPH, MGH
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FAST Lidocaine
Record Dates: First submitted 2006-10-11; First posted 2006-10-13 (Estimated); Last update posted 2009-02-26 (Estimated); Status verified 2009-02

CONDITIONS: Wounds
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: functional microarray — functional microarray application

SUMMARY:
The study's aim is to determine whether use of a mechanical device can improve the timeliness of anesthesia provided by liposomal lidocaine cream. Liposomal lidocaine cream has historically come in the brandnames of ELA-Max and LMX, with either 4% or 5% lidocaine in the cream. In this protocol, the abbreviation LLC will be generally used to refer to the 4% concentration to be used in FAST Lidocaine. Regardless of the concentration used, the encapsulation of lidocaine in liposomes protects the anesthetic from rapid metabolism and allows the medication to remain in the epidermis, yielding a theoretical benefit of long-lasting anesthesia.1 The test device is a painless functional microarray (FMA) that renders hundreds of microscopic punctures per cm2 in a patient's stratum corneum. The holes in the stratum corneum subsequently allow for faster movement of LLC into the skin to be anesthetized.

Currently, topical anesthetics are used less commonly in the Emergency Department (ED) than would be the case if the available approaches were not associated with such long onset times. The most commonly utilized topical anesthetic for intact skin, eutectic mixture of local anesthetics (EMLA), requires at least an hour for anesthetic effect; maximal effect requires up to 2 hours.2, 3 4 The topical anesthetic to be used in the FAST Lidocaine study, 4% LLC, has a roughly equipotent analgesic effect to that of EMLA and works faster, but must still be in place for at least a half-hour before onset of reliable anesthesia.1, 5-8 Commentators have judged such delays "considerable" and written that because of long application times, use of topical anesthetics may not be practical.1, 8-10 In discussing agents (such as LLC) that are formulated for more rapid transcutaneous absorption, ED wound care experts have written that "their delayed onset limits their use in the emergent setting."11 It has also been noted that LLC's utility is potentially diminished by the fact that anesthesia may begin to wear off as soon as 10 minutes after cream removal.8 Given the previously outlined findings, it is obvious that there is room for improvement in ED delivery of topical anesthesia. The goal of rendering topical anesthesia practical - and thus more likely to be used - constitutes the basis for the FAST Lidocaine study. We seek to identify whether a novel approach safely and painlessly improves the onset time (and perhaps depth) of topical anesthesia.

Reducing pain caused by procedures involving violation of the skin barrier (e.g. intravenous [IV] line placement, anesthesia and suturing of wounds) is an important goal. Needlesticks and IV catheters have been identified as important causes of pain in both children and adults.8, 12, 13 In terms of frequency, U.S. EDs place over 20 million IV catheters and care for over 10 million wounds.9 Thus, there is potentially broad-based utility in a potentiator for local anesthesia absorption in the ED.

The importance of the clinical goal of improving absorption of topical anesthesia has already prompted efforts aimed at improving delivery and efficacy of topically applied local anesthetics. Previous investigations have demonstrated utility - and limitations - of various methods of traversing and/or stripping the stratum corneum. Among the techniques studied have been use of electrical energy (iontophoresis),14 sound waves (sonophoresis),15, 16 adhesive tape17-19 and lasers.11, 12, 20, 21 While these varying approaches all have promise, their limitations leave room for assessment of a new method if it promises to be safe, painless, and effective.

The approach of the FAST Lidocaine study will be to assess FMA use. The FMA is a painless mechanism that is placed on the skin with minimal pressure. It creates microscopic punctures in the stratum corneum, facilitating movement of anesthetic through the cutaneous barrier. The device's physical characteristics, namely its easy application and low apparent potential for incorrect or unsafe use, appear quite suitable for ED utilization. If it works, the FMA would be immediately useful in a variety of circumstances.

The overarching goal of the FAST Lidocaine investigators is to assess whether the FMA can improve management of procedure-related pain in the ED. The main problem in terms of ED use of the currently available topical anesthetics - whether EMLA, LMX, or others - is the time of onset, rather than anesthetic efficacy. Thus, it is the timing impracticality for most ED situations that is the spur for FAST Lidocaine. The study's primary focus and endpoint will be time to anesthesia. Secondary analysis will evaluate whether the depth of anesthesia is improved by assessing the nadir of visual analog scale (VAS) assessments. However, it is noteworthy that deeper anesthesia is not necessary in order to establish the potential utility of FMA in the acute care setting.

ELIGIBILITY:
Inclusion Criteria:

* adults

Exclusion Criteria:

* no allergy to lidocaine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
anesthesia | hours

CONTACTS AND LOCATIONS:
Overall Officials: Stephen H Thomas, MD MPH, Principal Investigator — Massachusetts General Hospital